CLINICAL TRIAL: NCT01968915
Title: A Phase I Study of Oral LCL161 in Japanese Adult Patients With Advanced Solid Tumors
Brief Title: Safety and Tolerability of Oral LCL161 in Japanese Adult Patients With Advanced Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CLCL161A1102
Record Dates: First submitted 2013-10-21; First posted 2013-10-24 (Estimated); Last update posted 2020-12-19 (Actual); Status verified 2016-01

CONDITIONS: Neoplasms
Keywords: LCL161, Paclitaxel, Japanese patient, Neoplasms
MeSH Terms: conditions — Neoplasms | interventions — LCL161; Paclitaxel

ARMS (1):
- LCL161 (Experimental): Dose escalation part: Eligible patients will start to receive oral LCL161 once a week and will receive weekly paclitaxel, at 80 mg/m2 intravenous infusion over 1 hour, in combination with LCL161 from cycle 2. Dose expansion part: Eligible patients will receive oral LCL161 at the maximum tolerated dose and/or recommended dose in combination with weekly paclitaxel, at 80 mg/m2 intravenous infusion over 1 hour from cycle 1.
  Interventions: Drug: LCL161; Drug: Paclitaxel

INTERVENTIONS:
Drug: LCL161 — Patients will receive oral LCL161 once a week until unacceptable toxicity, disease progression and/or withdrawal of consent.
Drug: Paclitaxel — Patients will receive weekly paclitaxel as intravenous infusion over 1 hour in combination with LCL161, from cycle 2 in dose escalation part or from the first cycle in dose expansion part, and will continue it until unacceptable toxicity, disease progression and/or withdrawal of consent.

SUMMARY:
This study will evaluate safety and tolerability to estimate the maximum tolerated dose and/or recommended dose of oral LCL161 in Japanese patients with advanced solid tumors.

ELIGIBILITY:
Inclusion criteria:

1. Patients with a histologically or cytologically confirmed diagnosis of a solid tumor for which no further effective standard treatment is available.
2. ECOG performance status 0-1.
3. Patients must have recovered from all toxicities related to their previous treatment.

Exclusion criteria:

1. Unresolved nausea, vomiting, diarrhea or peripheral neuropathy CTCAE grade >1.
2. History of or current interstitial lung disease or autoimmune disease.
3. History of or current impaired cardiac function or clinically significant cardiac diseases.
4. Women of child-bearing potential, unless they are using highly effective methods of contraception.

Other protocol-defined inclusion/exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2013-11; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Frequency of dose limiting toxicities as a function of LCL161 during first cycle | First cycle (21 days)
Adverse events of oral LCL161 | From informed consent until 28 days after end of treatment (end of treatment visit occurs within 7 days after the determination of study discontinuation)
  Type and frequency of adverse events of oral LCL161 when administered in combination with weekly paclitaxel

SECONDARY OUTCOMES:
Adverse events of oral LCL161 | From informed consent until 28 days after end of treatment (end of treatment visit occurs within 7 days after the determination of study discontinuation)
  Type and frequency of adverse events of oral LCL161
LCL161 plasma concentration and derived pharmacokinetic parameters | From first cycle and up to 3 cycle (each cycle is 21-day period)
Paclitaxel plasma concentration and derived pharmacokinetic parameters | From first cycle of combination and up to 2 cycle (each cycle is 21-day period)
Tumor response according to RECIST 1.1 | Every 2 cycles for first 8 cycles, then every 3 cycles and until end of treatment (each cycle is 21-day period and end of treatment visit occurs within 7 days after the determination of study discontinuation)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (2):
- Japan (2):
  - Novartis Investigative Site, Nagoya, Aichi-ken
  - Novartis Investigative Site, Kobe, Hyōgo

REFERENCES:
- See also: Results for CLCL161A1102 can be found on the Novartis Clinical Trial Results Website — https://www.novctrd.com/ctrdweb/trialresult/trialresults/pdf?trialResultId=14605